CLINICAL TRIAL: NCT04031950
Title: Clinical Evaluation of a Paediatric Sleep Diagnosis Technology
Status: Recruiting | Type: Observational
Sponsor: Acurable Ltd. (Industry)
Collaborators: Sheffield Children's NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 269747
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- test group: Test group will wear PSG
  Interventions: Device: Novel wearable paediatric device
- Novel wearable device: THis group will wear the novel device
  Interventions: Device: Novel wearable paediatric device

INTERVENTIONS:
Device: Novel wearable paediatric device — The patient will wear the novel wearable paediatric device at the same time as polysmnography

SUMMARY:
The objective of this project is to gather research data and subsequently evaluate algorithms to demonstrate clinical efficacy of a novel sleep apnoea detection system in the paediatric population.

The Study will involve patients who will have been referred for diagnosis of sleep apnoea, and the ultimate aim will be to compare the output of a novel apnoea detection system against in -clinic polysomnography.

DETAILED DESCRIPTION:
The objective of this project is to gather research data and subsequently evaluate algorithms to demonstrate clinical efficacy of a novel sleep apnoea detection system in the paediatric population.

The Study will involve patients who will have been referred for diagnosis of sleep apnoea, and the ultimate aim will be to compare the output of a novel apnoea detection system against in -clinic polysomnography.

Patients who are referred to the clinic will spend one night's sleep in the clinic. They will wear a polysomnography system (current goldstandard) and the novel device.

At the end of the trial, we will compare the diagnosis results from both systems.

ELIGIBILITY:
Inclusion Criteria:

* Children older than one year old
* Children who have been referred to a sleep clinic due to suspicion of sleep apnoea.

Exclusion Criteria:

* Patients whose parents/legal guardians/carers are not fluent in English, or who have special communication needs.
* Known allergy to the adhesive dressing.
* Patients with physical or mental impairments who would be too distressed with additional sensors on themselves.
* Patients with not enough space on the neck area to fit the sensor.
* Clinical problem in the area in which the device will be attached, eg skin condition

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all children who have been referred for a sleep test.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Specificity and sensitivity of novel device | 6 months
  specificity and sensitivity of the output of the novel wearable device against polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Kingshott, PhD, Study Director — Sheffield Children's NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Sheffield Children Hospital, Sheffield
  - Southampton Children's Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No